CLINICAL TRIAL: NCT00160017
Title: Effectiveness and Cost-effectiveness of the Diabetes Integrated Care Breakthrough Collaborative to Improve Diabetes Care, Its Health Outcomes and Economic Costs
Brief Title: Effectiveness and Cost-effectiveness of the Diabetes Integrated Care Breakthrough Collaborative
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Dutch Institute for HealthCare Improvement (CBO) (Unknown); College of Health Insurances CVZ (Unknown)
Other Study IDs: Breakthrough_LoesSchouten; ZonMw grant no. 945-14-405
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
Keywords: Quality assurance health care; Diabetes; Breakthrough collaborative (IHI); Evaluation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- Collaborative group: Participants (i.e. profesionals) participate in a Breakthrough Collaborative intervention to improve diabetes care so that patients are provided more often with diabetes care as described in guidelines
  Interventions: Behavioral: Breakthrough collaborative
- usual care group: Participants are offered no intervention and care is provided as usual

INTERVENTIONS:
Behavioral: Breakthrough collaborative — Participants (professionals) participate in a Breakthrough Collaborative to improve diabetes care
  Groups: Collaborative group

SUMMARY:
The study tests whether implementing professional evidence-based guidelines and best practices for diabetes care -through participation of multidisciplinary teams in a Breakthrough collaborative- results in an improvement of diabetes care, its health outcomes and economic costs. Determinants of success are studied. Data on diabetes will also be used to better understand Breakthrough as an implementation or improvement method.

DETAILED DESCRIPTION:
Diabetes mellitus as a chronic disease is a major and growing health care problem. Studies on the prevention of severe complications provide evidence for the necessity of tight control. Different interventions and models to achieve strict control and reduce diabetes related risks of complications are available. These are, however, not implemented in daily practice. Our study focuses on this implementation problem: it tests whether implementing professional evidence-based guidelines and best practices -through participation of multidisciplinary teams in the Breakthrough collaborative- results in an improvement of diabetes care, its health outcomes and economic costs.

Data on diabetes will also be used to explore and better understand the Breakthrough model as an implementation method. Only uncontrolled observational studies have, so far, described the outcomes of Breakthrough collaboratives. They also describe significant differences between teams in specific improvements made in patient care and organisational performance, resulting in different implementation and medical costs. There is hardly any information regarding these costs and the cost-effectiveness of collaboratives, and little knowledge about how they could be made more effective. Insight is also needed into the factors that influence the success of individual teams. There are no data regarding the sustainability of improvements.

ELIGIBILITY:
Inclusion Criteria:

* each patient, male or female, visiting the hospital outpatient clinic or general practice with type II diabetes mellitus during a specified period. Patients should be able to read and write the Dutch language.

Exclusion Criteria:

* pregnancy
* patients with a life expectancy < 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 6 intervention and 9 control sites representing multiporfessional provider teams from 13 outpatient clinics (47 internists) and 37 general practices (42 general practitioners)
  NB To assess the effects of the collaborative, patient outcomes, professional performance, and structural aspects of care management are measured. Patients visiting the clinics were invited to participate by filling out questionnaires and providing written consent to have their medical records examined. Below information on patient inclusion is provided.
Sampling Method: Non-Probability Sample
Enrollment: 1861 (Actual)
Dates: Start 2005-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
HbA1c | baseline, after 12 months and after 24 months

SECONDARY OUTCOMES:
To improve the patient outcomes mentioned above, teams are supported: | baseline, after 12 months and after 24 months
(I) to introduce self-management of patients, | baseline, after 12 months and after 24 months
(II) to change professional performance and the organisation of care (by implementing guidelines and local protocols focusing on the prevention of severe complications and introducing diabetes nurses) and | baseline, after 12 months and after 24 months
(III) to introduce a system to administrate clinical parameters. | baseline, after 12 months and after 24 months
These intermediate outcomes will be measured as well, in both the intervention and the control group. | baseline, after 12 months and after 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Marlies E.J.L. Hulscher, MSc, PhD, Principal Investigator — Radboud University Nijmegen Medical Centre, Centre for Quality of Care Research; Louis W. Niessen, MD, PhD, Principal Investigator — Erasmus Institute for Medical Technology Assessment, Institute of Health Policy and Management (iBMG); Richard PTM Grol, Prof., Study Director — Radboud University Nijmegen Medical Centre, Centre for Quality of Care Research; Robbert Huijsman, Prof., Study Director — Erasmus Institute for Medical Technology Assessment, Institute of Health Policy and Management (iBMG)
Locations (52):
- Netherlands (52):
  - Universitair Medisch Centrum St Radboud, Nijmegen, Gelderland
  - Huisartspraktijk28, Nijmegen, Gelderland
  - Atrium Medisch Centrum, Polikliniek Interne Geneeskunde, Kerkrade, Limburg
  - Huisartsenpraktijk Julianastraat14, Asten, North Brabant
  - Huisartspraktijk De Poort10, Beuningen, North Brabant
  - Praktijk Van Mechelen32, Dinteloord, North Brabant
  - Huisartspraktijk33, Fijnaart, North Brabant
  - St. Annaziekenhuis, Maatschap Interne Geneeskunde, Geldrop, North Brabant
  - Huisartsenpraktijk Scholten17, Helmond, North Brabant
  - Huisartsenpraktijk Dams15, Helmond, North Brabant
  - Quartz Transmuraal Centrum voor de Regio Helmond, Elkerliek ziekenhuis Provisorium 1e etage, Helmond, North Brabant
  - Huisartsenpraktijk van den Nieuwenhof16, Helmond, North Brabant
  - Huisartspraktijk34, Roosendaal, North Brabant
  - Huisartspraktijk31, Roosendaal, North Brabant
  - Huisartspraktijk13, Roosendaal, North Brabant
  - Huisartspraktijk Vincenten12, Roosendaal, North Brabant
  - Huisartspraktijk30, Roosendaal, North Brabant
  - Huisartspraktijk22, Someren, North Brabant
  - Artsenpraktijk Ruiterstal11, Steenbergen, North Brabant
  - Huisartspraktijk De Heelhoek9, Wijchen, North Brabant
  - Medisch Centrum Alkmaar, Alkmaar, North Holland
  - Huisartspraktijk1, Alkmaar, North Holland
  - Huisartspraktijk24, Amsterdam, North Holland
  - St. Lucas Andreas Ziekenhuis, Amsterdam, North Holland
  - Huisartspraktijk29, Amsterdam, North Holland
  - Slotervaartziekenhuis, Maatschap Interne, Amsterdam, North Holland
  - Huisartspraktijk18, Amsterdam, North Holland
  - Huisartspraktijk20, Amsterdam, North Holland
  - Huisartspraktijk19, Amsterdam, North Holland
  - Onze Lieve Vrouwe Gasthuis, Amsterdam, North Holland
  - Huisartspraktijk21, Amsterdam, North Holland
  - Huisartspraktijk23, Amsterdam, North Holland
  - Huisartspraktijk25, Amsterdam, North Holland
  - Huisartspraktijk5, Den Helder, North Holland
  - Gemini Ziekenhuis, Den Helder, North Holland
  - Gezondheidscentrum "De Schooten"6, Den Helder, North Holland
  - Spaarne Ziekenhuis, Afdeling Inwendige Geneeskunde, Haarlem, North Holland
  - Huisartspraktijk27, Limmen, North Holland
  - Huisartspraktijk26, Schoorl, North Holland
  - Therapeuticum Lemminkäinen36, Groningen, Provincie Groningen
  - Academisch Ziekenhuis Groningen, Afdeling Inwendige Geneeskunde, Groningen, Provincie Groningen
  - Huisartspraktijk35, Groningen, Provincie Groningen
  - Huisartspraktijk7, Zuidhorn, Provincie Groningen
  - Huisartspraktijk2, Hoofddorp, South Holland
  - Huisartspraktijk3, Hoofddorp, South Holland
  - Medisch Centrum Het Joppe8, Leiden, South Holland
  - Gezondheidscentrum Stevenshof4, Leiden, South Holland
  - Leids Universitair Medisch Centrum, Leiden, South Holland
  - Diaconessenhuis, Leiden, South Holland
  - Mesos Medisch Centrum, Bilthoven, Utrecht
  - Gezondheidscentrum Kanaleneiland38, Utrecht, Utrecht
  - Huisartspraktijk Carnegiedreef37, Utrecht, Utrecht

REFERENCES:
- [Derived] Schouten LM, Niessen LW, van de Pas JW, Grol RP, Hulscher ME. Cost-effectiveness of a quality improvement collaborative focusing on patients with diabetes. Med Care. 2010 Oct;48(10):884-91. doi: 10.1097/MLR.0b013e3181eb318f. PMID 20808258
- See also: Information about the Centre for Quality of Care Research — http://www.wokresearch.nl